CLINICAL TRIAL: NCT03083509
Title: A Physiological Profile of Recovery From Mechanical, Metabolic, and Mixed Exercise Stressors
Brief Title: A Physiological Profile of Recovery From Resistance, Endurance, and Mixed Exercise Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 205085
Record Dates: First submitted 2016-09-28; First posted 2017-03-20 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Sports Nutritional Sciences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group1 (Resistance trained individuals) (Other): Resistance trained individuals (>3 sessions per weeks for ≥2 years with a minimum of 1 session per week including leg-based exercises)
  Interventions: Other: Resistance exercise weight training session
- Group 2 (Trained cyclists) (Other): Trained cyclists (competing at a minimum of Category 3 road racing/estimated 10 mile TT of <25 minutes and a training history of ≥5 hours per week for ≥2 years)
  Interventions: Other: High-Intensity stochastic cycling session
- Group 3 (Team sports players) (Other): Team sports players (minimum of University 1st team level e.g. soccer, rugby union, rugby league, hockey and basketball, playing competitively ≥1x per week for ≥2 years)
  Interventions: Other: Simulated Team sport protocol

INTERVENTIONS:
Other: Resistance exercise weight training session — A resistance exercise session was performed. Following a warm-up that consisted of five-minutes cycling at a self-selected intensity, as well as three progressive lifts at 50, 75, and 90% 6 rep max (RM), participants performed four sets of six repetitions at 100% of 6RM (as determined by the maximal weight lifted during the maximal strength assessment) of the following lifts; back squat, front squat, good mornings, and Bulgarian split-squat. Two minutes rest was afforded between sets and exercises.
  Arms: Group1 (Resistance trained individuals)
Other: High-Intensity stochastic cycling session — A high-intensity stochastic cycling session was performed. The cycling protocol was performed using a magnetically-braked cycle ergometer (Velotron, RacerMate). Following a 10 minute standardised warm-up including 3 × 3s sprints, participants completed a simulated road-race, consisting of sprints of varied length, differing work to rest ratios and short time-trials.
  Arms: Group 2 (Trained cyclists)
Other: Simulated Team sport protocol — A simulated team sport protocol was performed. Participants performed a standardised warm-up consisting of performing three laps of the circuit jogging, and three laps at 50, 75, and 90% of perceived maximal speed. Participants were then afforded five minutes to perform self-selected stretching prior to commencing the session. Participants performed two sets of 45 minutes of the simulated team sport protocol, separated by 15 minutes rest. Each 45 minute period consisted of a one minute circuit repeated 45 times that replicates typical movement patterns observed during team sports and includes walking, jogging, jumping, sprinting, agility, and decelerations. Each circuit was initiated on the minute, therefore enabling participants to rest following the completion of each circuit. Pilot testing showed participants completes each circuit in approximately 48-55 seconds (sec) therefore enabling 5-12sec rest after each circuit.
  Arms: Group 3 (Team sports players)

SUMMARY:
The aim of this study to increase understanding of physiological and functional perturbations following a continuum of exercise stressors.

DETAILED DESCRIPTION:
This study utilised a between groups design, with a within-groups control. This allowed the within-subject profiling of recovery during both a control and exercise week. This design also allowed each group to perform an ecologically valid exercise session as well as having markers of recovery tailored to the areas of interest specific to each cohort. By having each group perform a non-exercise control week, this gives valuable information on the reliability and smallest worthwhile change for a range of both novel and commonly used recovery markers.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent (see Appendices 2-4) and has received a signed and dated copy of the informed consent form.
* Participant is male
* Good general and mental health as assessed by a health questionnaire and with, in the opinion of the investigator or medically qualified designee ,no clinically significant and relevant abnormalities in medical history or upon oral examination. As well as absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* Participants will be fully briefed prior to agreeing to participate in the study and the research team will confirm that they are willing, able, and likely to comply with all procedures and complete the study.
* Only the following individuals will be recruited as participants for the study:

Group 1: Resistance trained individuals (≥3 sessions per week for ≥2 years with a minimum of 1 session per week including leg-based exercises).

Group 2: Trained cyclists (competing at a minimum of Category 3 roadracing/ estimated 10 mile TT of <25 minutes and a training history of ≥5 hours per week for ≥2 years).

Group 3: Team sports players (minimum of University 1st team level e.g. soccer, rugby union, rugby league, hockey, and basketball, playing competitively ≥1x per week for ≥2 years).

Exclusion Criteria:

* Individuals that do not fit the training status inclusion criteria.
* Current use of any non-steroidal anti-inflammatory drugs (NSAID's) or other analgesics for pain relief.
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last 1 year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* Have a heart or any other medical condition that may contra-indicate participants from taking part in high intensity or exhaustive physical activity.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
Maximal isometric volume contraction (MIVC) | Up to Day 26
  Following a five minute warm-up cycling at 100W (Power output of the cycle in watts), participants seated on a dynamometer. For each participant the chair height, length and dynamometer position were recorded and maintained in subsequent trials. Participants completed a standardised warm-up consisting of contractions at 50, 75, and 90% of perceived maximal force. Participants then performed three MIVC of the dominant limb each lasting approximately 3 seconds (sec). Sixty seconds rest was given in between repetitions with peak force (N) recorded and the best attempt used for subsequent analysis.
Rate of force development (RFD) | Up to Day 26
  Participants were instructed to stand with their feet approximately shoulder width apart on a force plate, with hands placed on hips. Participants completed a standardised warm-up consisting of jumps at 50, 75, and 90% of perceived maximum jump height. Participants were instructed to perform a maximal vertical jump by using their own choice of depth and pace (whilst maintaining hands on hips throughout) and to land with straight legs. If flight time is exaggerated by participants removing hands from the hips or bending their legs whilst in the air, the test was performed again. Three maximal efforts were performed with sixty seconds rest in between repetitions, RFD (N·s-1) recorded, and the best attempt used for subsequent analysis.
Countermovement jump (CMJ) | Up to Day 26
  Participants were instructed to stand with their feet approximately shoulder width apart on a force plate, with hands placed on hips. Participants completed a standardised warm-up consisting of jumps at 50, 75, and 90% of perceived maximum jump height. Participants were instructed to perform a maximal vertical jump by using their own choice of depth and pace (whilst maintaining hands on hips throughout) and to land with straight legs. If flight time is exaggerated by participants removing hands from the hips or bending their legs whilst in the air, the test was performed again. Three maximal efforts were performed with sixty seconds rest in between repetitions with jump height (cm) recorded, and the best attempt was used for subsequent analysis.
20 meter (m) sprint assessment (Group 1 and 3 only) | Up to Day 26
  A 20 m runway in an indoor track was marked using cones and two sets of infrared timing gates, one set at each end of the start and finish line. Participants completed a standardised warm-up consisting of performing 20 m runs at 50, 75, and 90% of perceived maximal effort. Participants stand 0.3 m behind the start line to avoid premature triggering of the timing system, and were instructed to lead with the same starting leg for all attempts before performing three sprints interspersed with 60sec rest. Sprint time (sec) was recorded and the best attempt was used for subsequent analysis.
Cycling Time-Trial performance assessment (Group 2 only) | Up to Day 26
  Following a standardised five minute warm-up at 100 W, with a 10sec sprint at 2 minutes 30 sec, participants completed a 5 minute all-out time trial, covering as much distance as possible. Participants were initially instructed that they were to cover as much distance as possible in 5 minutes, before being blinded to time and test performance and informed of the half-way stage by the investigator. Distance covered (m), mean power (W) and work done (J) were calculated and used for subsequent analysis.

SECONDARY OUTCOMES:
Sleep efficiency | Up to Day 26
  Sleep efficiency was measured with a wrist-strap Actigraph worn at all the times by participants from Visits 3-7 and 8-12. Data from the Actigraph was uploaded to a secure cloud-based Web application and selected variable was used for subsequent analysis.
Sleep latency | Up to Day 26
  Sleep latency was measured with a wrist-strap Actigraph worn at all the times by participants from Visits 3-7 and 8-12. Data from the Actigraph was uploaded to a secure cloud-based Web application and selected variable was used for subsequent analysis.
Time in bed | Up to Day 26
  Time in bed was measured with a wrist-strap Actigraph worn at all the times by participants from Visits 3-7 and 8-12. Data from the Actigraph was uploaded to a secure cloud-based Web application and selected variables were used for subsequent analysis.
Time asleep | Up to Day 26
  Time asleep was measured with a wrist-strap Actigraph worn at all the times by participants from Visits 3-7 and 8-12. Data from the Actigraph was uploaded to a secure cloud-based Web application and selected variables were used for subsequent analysis.
Perceived muscle soreness | Up to Day 26
  Active muscle soreness was determined using a 200 millimeter (mm) visual analogue scale with "no pain" indicated at one end and "pain/soreness as bad as it could be" at the other. Participants stand with the hands on hips and feet approximately shoulder width apart. The participant then performed a squat to 90°, before standing and recording the pain felt in the lower limbs.
Perceived recovery measured by the daily analyses of life demands for athletes (DALDA) questionnaire | Up to Day 26
  DALDA questions were scored using following scale: worse than normal, Normal and Better than normal.
Interleukin 10 (IL-10) | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
Interleukin 6 (IL-6) | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
C-reactive protein | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
Neutrophils | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
Creatine kinase | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
F2-isoprostanes | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
Protein carbonyls | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
Fast myosin | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
Slow myosin | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
Matrix metalloproteinase-9 | Up to Day 26
  Venous blood samples were collected using the venipuncture technique from a vein in the ante-cubital fossa region by a trained phlebotomist. Two samples (2 × 5milileter [mL]) were collected per participant at visits 3 (×3), 4, 5, 6, 7, 8 (×3), 9, 10, 11, and 12. Visits 3-7 and 8-12 were separated by 24hours and will occur on consecutive days. During visits 3 and 8, samples were taken at baseline as well as 2h and 6h post control/exercise. Additionally on visits 3 (×3), 4, 5, 8 (×3), 9, and 10 a 2mL blood draw taken for 600uL of whole blood to be processed and stored at -80 degrees until further analysis for the quantification of GSH:GSSG ratio. Visits 7 and 8 were separated by approximately two weeks, therefore totaling a collection volume of 160mL blood over approximately a four week period. All Blood samples were analysed by enzyme-linked immunosorbent assay (ELISA) technique.
Limb Girth | Up to Day 26
  Lower limb girth was measured at the mid-thigh on the dominant leg. Mid-thigh was defined as the halfway point between the anterior superior iliac spine and the proximal aspect of the patella. All measurements were taken with the participant standing in anatomical zero with thigh muscles relaxed. A line semi permanently marked around the circumference of the dominant thigh to ensure the reliability of measurements between sessions. The mean of three measurements was used for subsequent analysis. The same investigator will record the measurements between sessions and intra-rater reliability will be reported
Range of motion (ROM) assessment | Up to Day 26
  A goniometer was used to measure the relaxed and flexed knee joint angles of the dominant limb. Measurements was taken when the participants maximally flexes the knee joint to touch the hip with the heel while keeping the knee joint at the side of the body in the anatomical zero position. Maximal extension was taken when the participant extends the knee joint as much as possible and was allowed to hold onto a wall for balance. The mean of three measurements was taken for flexion and extension and ROM was calculated by subtracting flexion from extension. The same investigator will record the measurements between sessions and intra-rater reliability was reported.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Brentford, United Kingdom

IPD SHARING:
Plan to Share IPD: No